CLINICAL TRIAL: NCT01700387
Title: A Randomized, Pilot Study to Evaluate the Tolerability of OnabotulinumtoxinA Plus Topiramate vs. OnabotulinumtoxinA Plus Placebo and Long Term Effect of Treatment on Cognitive Efficiency and Continuation of Care
Brief Title: A Study to Evaluate the Tolerability of Botox and Topiramate or Botox and Placebo and Effect on Cognitive Efficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-001AL; 71403 (Other Grant/Funding Number: Allergan)
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Chronic Migraine
Keywords: Migraine; Chronic Migraine; Cognitive Efficiency; Pilot Study; Long Term Effect
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OnabotulinumtoxinA + Topiramate (Experimental): Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with topiramate. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: topiramate 25 mg qhs Week 2: topiramate 25 mg bid Week 3: topiramate 25 mg q am + topiramate 50 mg qhs Week 4: topiramate 50 mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
  Interventions: Drug: onabotulinumtoxinA; Drug: Topiramate
- OnabotulinumtoxinA + Placebo (Placebo Comparator): Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with placebo. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: 1 tab qhs Week 2: 1 tab bid Week 3: 1 tab q am + 2 tabs qhs Week 4: 2 tabs bid
  Interventions: Drug: onabotulinumtoxinA; Drug: Placebo

INTERVENTIONS:
Drug: onabotulinumtoxinA — All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
  Other Names: Botox, Botulinum Toxin Type A Purified Neurotoxin Complex
Drug: Topiramate — Subjects randomized to the onabotulinumtoxinA + topiramate group will receive:
  Week 1: topiramate 25 mg qhs Week 2: topiramate 25 mg bid Week 3: topiramate 25 mg q am + topiramate 50 mg qhs Week 4: topiramate 50 mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
  Other Names: Topamax
  Arms: OnabotulinumtoxinA + Topiramate
Drug: Placebo — Subjects randomized to the onabotulinumtoxinA + placebo group will receive:
  Week 1: placebo 25 mg qhs Week 2: placebo 25 mg bid Week 3: placebo 25 mg q am + placebo 50 mg qhs Week 4: placebo 50 mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
  Arms: OnabotulinumtoxinA + Placebo

SUMMARY:
The purpose of this study is to evaluate sustained tolerability, quality of life, and change in cognitive efficiency following treatment with OnabotulinumtoxinA and daily topiramate vs. OnabotulinumtoxinA and daily placebo (Group A vs. Group B).

DETAILED DESCRIPTION:
Numerous migraine preventive medications are well known to be associated with cognitive impairment and disruption of mood.

Clinvest would propose a pilot study of chronic migraine patients randomized 1:1 to onabotulinumtoxinA and daily topiramate or onabotulinumtoxinA and placebo. This pilot study will examine the degree to which subjects are able to tolerate and are satisfied with a migraine preventive medication in addition to onabotulinumtoxinA over an extended period of time and the effect of the subjects' quality of life compared with onabotulinumtoxinA as a single therapy. It will also assess short and long term effects of these two treatments on cognition. Cognitive performance will be measured by the Mental Efficiency Workload Test (MEWT), a repeated measures handheld neuropsychological test battery that measures mental efficiency via 4 sub-tests (Simple Reaction Time, Running Memory, Continuous Performance Task, Matching to Sample, and Mathematical Processing) to demonstrate short and long term changes in mental status compared to their baseline. The Controlled Oral Word Association Test (COWAT) will be used to test verbal fluency and screen for anomic aphasia, a known side effect of several migraine prophylactic medications including topiramate.

Visit 1 - Screening / Baseline Following Informed Consent a medical, headache, and medication history will be collected and a physical and neurological exam performed on all subjects. A urine pregnancy test will be collected from any subject of child-bearing potential. Vital signs and ECG (at the discretion of the investigator) will be completed. The Mental Efficiency Workload Test (MEWT) will be administered 3 times to establish a cognitive efficiency baseline. The COWAT will be completed. Subjects will be instructed regarding completion of the online 1-month Baseline Period Migraine Diary and be instructed to treat headaches during the 1-month Baseline Period with their usual acute migraine medication in their usual manner.

Visit 2 - Randomization / Injection Following the 1-month Baseline Period, any change in medical or medication history since the previous visit will be collected and a pregnancy test collected if appropriate. Vital signs will be recorded. Subjects continuing to meet eligibility criteria will be instructed to complete the online Treatment Period Migraine Diary daily. The MEWT, HIT-6, Migraine Specific Questionnaire (MSQ) and COWAT will be completed. The coordinator will assess compliance with online headache diary and any deviation outside of 100% compliance should be documented at the site. If in the investigator's opinion, the subject maintained a high level of compliance with the online headache diary, subjects will then be randomized into the study.

Eligible subjects will be randomized 1:1 in a blinded fashion to receive onabotulinumtoxinA at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas and daily topiramate (Group A) or onabotulinumtoxinA at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas and placebo to match topiramate (Group B).

Daily study medication (topiramate or placebo) will be dispensed for the following 3 months.

The Group A topiramate titration schedule will be as follows:

Week 1: topiramate 25 mg qhs (every night at bedtime) Week 2: topiramate 25 mg bid (twice a day) Week 3: topiramate 25 mg q am (everyday before noon) + topiramate 50 mg qhs Week 4: topiramate 50mg bid

Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.

The Group B placebo schedule will be as following:

Week 1: 1 tab qhs Week 2: 1 tab bid Week 3: 1 tab q am + 2 tabs qhs Week 4: 2 tabs bid

Subjects will be instructed to complete the online daily Treatment Period Migraine Diary during the next 3-month period.

Following Visit 2, subjects will be phoned monthly and any adverse events collected. Subjects will also be sent weekly reminders for 8 weeks following Visit 2 via email to take study medication, complete online diary and contact their coordinator for any questions or concerns they may have. During the titration period, any subject in Group A experiencing an adverse event thought to be related to study medication dosage will return to the clinic at an Unscheduled Visit for dosage adjustment.

Visit 3

Three months following Visit 2, subjects will return and complete the MEWT, HIT-6, MSQ, COWAT, and Subject's Global Impression of Change (SGIC). The Investigator will complete a Physician's Global Impression of Change (PGIC). Any change in medical or medication history since the previous visit will be collected and a pregnancy test collected if appropriate. Vital signs will be recorded. The coordinator will assess compliance with online headache diary and any deviation outside of 100% compliance should be documented at the site. If in the investigator's opinion, the subject maintained a high level of compliance with the online headache diary, subjects will be allowed to continue in the study.

All subjects will be administered a dose of 155 U onabotulinumtoxinA at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas.

Any unused study medication and used packaging will be collected, drug accountability will be performed, and daily study medication (topiramate or placebo) will be dispensed for the following 3 months.

Subjects will be instructed to complete the online daily Treatment Period Migraine Diary during the next 3-month period.

Following Visit 3, subjects will be phoned monthly and any adverse events collected.

Visit 4

Three months following Visit 3, subjects will return and complete the MEWT, HIT-6, MSQ, COWAT, and Subject's Global Impression of Change (SGIC). The Investigator will complete a Physician's Global Impression of Change (PGIC). Any change in medical or medication history since the previous visit will be collected and a pregnancy test collected if appropriate. Vital signs will be recorded. The coordinator will assess compliance with online headache diary and any deviation outside of 100% compliance should be documented at the site.

All subjects will be administered a dose of 155 U onabotulinumtoxinA at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas.

Any unused study medication and used packaging will be collected, drug accountability will be performed, and daily study medication (topiramate or placebo) will be dispensed for the following 3 months.

Subjects will be instructed to complete the online daily Treatment Period Migraine Diary during the next 3-month period.

Following Visit 4, subjects will be phoned monthly and any adverse events collected.

Visit 5

Three months following Visit 4, subjects will return and complete the MEWT, HIT-6, MSQ, COWAT, and Subject's Global Impression of Change (SGIC). The Investigator will complete a Physician's Global Impression of Change (PGIC). Any change in medical or medication history since the previous visit will be collected and a pregnancy test collected if appropriate. Vital signs will be recorded. The coordinator will assess compliance with online headache diary and any deviation outside of 100% compliance should be documented at the site.

All subjects will be administered a dose of 155 U onabotulinumtoxinA at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas.

Any unused study medication and used packaging will be collected, drug accountability will be performed, and daily study medication (topiramate or placebo) will be dispensed for the following 3 months.

Subjects will be instructed to complete the online daily Treatment Period Migraine Diary during the next 3-month period.

Following Visit 5, subjects will be phoned monthly and any adverse events collected.

Visit 6

Three months following Visit 5, subjects will return and complete the MEWT, HIT-6, MSQ, COWAT, and Subject's Global Impression of Change. The Investigator will complete a Physician's Global Impression of Change. Any change in medical or medication history since the previous visit will be collected and a pregnancy test collected if appropriate. Vital signs will be recorded. The coordinator will assess compliance with online headache diary and any deviation outside of 100% compliance should be documented at the site.

Any unused study medication and used packaging will be collected and drug accountability will be performed.

Subjects will exit the study at Visit 6.

ELIGIBILITY:
Inclusion Criteria:

1. must be outpatient, male or female, of any race, between 18 and 65 years of age.
2. if female of child bearing potential must have a negative pregnancy test result at the Screening Visit and practice a reliable method of contraception.

   A female is considered of childbearing potential unless she is post-menopausal for at least 12 months prior to administration of study drug, without a uterus and/or both ovaries or has been surgically sterilized for at least 6 months prior to study drug administration.

   Reliable methods of contraception are:

   Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product. Throughout the study, and for a time interval (5 days) after completion or premature discontinuation from the study. History of bilateral tubal ligation Sterilization of male partner; or, Implants of levonorgestrel; or, Injectable progestogen, or, Oral contraceptive (combination therapy with ethinyl estradiol plus a progestin) with a placebo week every 1-3 months; or, Any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year (not all IUD's meet this criterion) in use at least 30 days prior to study drug administration; or, Spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm); or, Any other barrier methods (only is used in combination with any of the above acceptable methods) in use at least 14 days prior to study drug administration; or, Any other methods with published data showing that the highest expected failure rate for that method is less than 1% per year.
3. must have history of chronic migraine (with or without aura) according to the criteria proposed by the Headache Classification Committee of the International Headache Society (IHS) for at least 3 months prior to enrollment.
4. must be able to understand the requirements of the study including maintaining a headache Diary, and signing informed consent.
5. must be in good general health as determined by investigator.
6. if taking migraine preventive, must be on a stable dose of preventive medication for at least 6 weeks prior to screening.
7. must have daily access to internet for completion of online daily headache diary.

Exclusion Criteria:

1. if female, is pregnant, planning to become pregnant during the study period, are breast feeding, or are of childbearing potential and not practicing a reliable form of birth control.
2. has headache disorders outside IHS-defined chronic migraine definition.
3. has evidence of underlying pathology contributing to their headaches.
4. has any medical condition that may increase their risk with exposure to OnabotulinumtoxinA including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function.
5. has profound atrophy or weakness of muscles in the target areas of injection.
6. has skin conditions or infections at any injection site.
7. has allergy or sensitivities to any component of the test medication.
8. has previously received onabotulinumtoxinA for migraine prevention.
9. has previously received topiramate.
10. who in the opinion of the investigator, has active major psychiatric or depressive disorders including alcohol/drug abuse.
11. meets International Headache Society criteria for Medication Overuse Headache with opioid or butalbital containing products.
12. who in the opinion of the investigator, is taking opioid or butalbital containing products more than once a week that could be contributing to a pattern of increased headaches or cognitive decline.
13. is planning or requiring surgery during the study.
14. has a history of poor compliance with medical treatment.
15. is currently participating in an investigational drug study or has participated in an investigational drug study within the previous 30 days of the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (1):
- Clinvest/A Division of Banyan Group, Inc., Springfield, Missouri, United States

REFERENCES:
- [Result] Bootsma HP, Aldenkamp AP, Diepman L, Hulsman J, Lambrechts D, Leenen L, Majoie M, Schellekens A, de Krom M. The Effect of Antiepileptic Drugs on Cognition: Patient Perceived Cognitive Problems of Topiramate versus Levetiracetam in Clinical Practice. Epilepsia. 2006;47 Suppl 2:24-7. doi: 10.1111/j.1528-1167.2006.00683.x. PMID 17105455
- [Result] Kim SY, Lee HW, Jung DK, Suh CK, Park SP. Cognitive Effects of Low-dose Topiramate Compared with Oxcarbazepine in Epilepsy Patients. J Clin Neurol. 2006 Jun;2(2):126-33. doi: 10.3988/jcn.2006.2.2.126. Epub 2006 Jun 20. PMID 20396496
- [Result] Meador KJ, Loring DW, Vahle VJ, Ray PG, Werz MA, Fessler AJ, Ogrocki P, Schoenberg MR, Miller JM, Kustra RP. Cognitive and behavioral effects of lamotrigine and topiramate in healthy volunteers. Neurology. 2005 Jun 28;64(12):2108-14. doi: 10.1212/01.WNL.0000165994.46777.BE. PMID 15985582

RESULTS

PARTICIPANT FLOW:
Groups:
- OnabotulinumtoxinA + Topiramate: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with topiramate. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: topiramate 25 mg qhs (every night at bedtime) Week 2: topiramate 25 mg bid (twice a day) Week 3: topiramate 25 mg q am (every day before noon) + topiramate 50 mg qhs Week 4: topiramate 50 mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
- OnabotulinumtoxinA + Placebo: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with placebo. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: 1 tab qhs (every night at bedtime) Week 2: 1 tab bid (twice daily) Week 3: 1 tab q am (every day before noon) + 2 tabs qhs Week 4: 2 tabs bid
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
Period: Overall Study
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Started | 10 | 10
Completed | 6 | 6
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Only those subjects which randomized were included in the baseline analysis.
Groups:
- OnabotulinumtoxinA + Topiramate: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with topiramate. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: topiramate 25 mg qhs Week 2: topiramate 25 mg bid Week 3: topiramate 25 mg q am + topiramate 50 mg qhs Week 4: topiramate 50 mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
- OnabotulinumtoxinA + Placebo: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with placebo. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: 1 tab qhs Week 2: 1 tab bid Week 3: 1 tab q am + 2 tabs qhs Week 4: 2 tabs bid
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.84 (15.98) | 39.51 (6.99) | 40.18 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Subject Attrition Post Randomization
Description: Count of subject attrition following randomization and reason for attrition (Consent withdrawn, Withdrawn due to adverse event, Lost to follow up)
Time Frame: Collected on Visit 2 (Day 29) through Visit 6 (Day 365)
Measure: Number; unit: participants
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 10 | 10
participants
  Consent Withdrawn | 1 | 2
  Withdrawn Due to Adverse Event | 1 | 1
  Lost to Follow Up | 2 | 1

2. Primary Outcome: Subject Global Impression of Change (SGIC)
Description: Score on Subject Global Impression of Change at Visits 3-6 (Day 113 and 365). Likert scale ranging from 1-7, where 1 = extremely worse and 7 = extremely better.
Time Frame: Collected on Visit 3 (Day 113), Visit 4 (Day 197), Visit 5 (281), and Visit 6 (Day 365)
Population: Number of participants vary at each visit based on the number of those still enrolled in the study at the time of the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OnabotulinumtoxinA + Topiramate: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with topiramate. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: topiramate 25 mg q hs Week 2: topiramate 25 mg bid Week 3: topiramate 25 mg q am + topiramate 50mg q hs Week 4: topiramate 50mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
- OnabotulinumtoxinA + Placebo: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with placebo. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: 1 tab q hs Week 2: 1 tab bid Week 3: 1 tab q am + 2 tabs q hs Week 4: 2 tabs bid
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 8 | 10
units on a scale
  Visit 3 | 5.38 (1.19) | 5.30 (1.25)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | 6.33 (0.82) | 5.77 (1.09)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | 6.66 (0.52) | 6.17 (1.17)
  Visit 6: number analyzed (Participants) | 6 | 6
  Visit 6 | 7.00 (0.00) | 6.00 (1.26)

3. Primary Outcome: Physician Global Impression of Change (PGIC)
Description: Score on Physician Global Impression of Change at Visits 3-6 (Day 113 and 365). Likert scale ranging from 1-7, where 1 = extremely worse and 7 = extremely better.
Time Frame: Collected on Visit 3 (Day 113), Visit 4 (Day 197), Visit 5 (281), and Visit 6 (Day 365)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 8 | 10
units on a scale
  Visit 3 | 5.25 (1.16) | 5.30 (1.25)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | 5.40 (1.34) | 5.89 (0.93)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | 6.67 (0.52) | 5.83 (1.94)
  Visit 6: number analyzed (Participants) | 6 | 6
  Visit 6 | 6.83 (0.41) | 5.83 (1.47)

4. Primary Outcome: Subject's Controlled Oral Word Association Test (COWAT) Score Percent Change Compared From Baseline to Visits 3-6
Description: The Controlled Oral Word Association Test (COWAT) is a measure of verbal fluency. Raw COWAT scores have a lower bound of 0 with no upper bound. Higher scores indicate better verbal fluency. COWAT score percent change from baseline will be reported. Positive change scores represent better verbal fluency compared to baseline.
Time Frame: Baseline, Visit 3 (Day 113) through Visit 6 (Day 365)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline score
Groups:
- OnabotulinumtoxinA + Topiramate: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with topiramate. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: topiramate 25 mg qhs Week 2: topiramate 25 mg bid Week 3: topiramate 25 mg q am + topiramate 50 mg qhs Week 4: topiramate 50 mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
  Topiramate: Subjects randomized to the onabotulinumtoxinA + topiramate group will receive:
  Week 1: topiramate 25 mg qhs Week 2: topiramate 25 mg bid Week 3: topiramate
- OnabotulinumtoxinA + Placebo: Subject will receive 155 U onabotulinumtoxinA injections at 31 sites every 3 months for 12 months and treat daily with placebo. During the first month of the treatment period, subjects will titrate as follows:
  Week 1: 1 tab qhs Week 2: 1 tab bid Week 3: 1 tab q am + 2 tabs qhs Week 4: 2 tabs bid
  onabotulinumtoxinA: All subjects will receive a minimum dose of 155 U Botulinum Toxin Type A Purified Neurotoxin Complex administered at 31 fixed-site, fixed-dose injections across seven (7) specific head/neck muscle areas at Visits 2-5.
  Placebo: Subjects randomized to the onabotulinumtoxinA + placebo group will receive:
  Week 1: placebo 25 mg qhs Week 2: placebo 25 mg bid Week 3: placebo 25 mg q am + placebo 50 mg qhs Week 4: placebo 50 mg bid Only one dosage adjustment (increase or decrease), based on efficacy or tolerability, may be made at the investigator's discretion. Subjects must maintain a dose of at least 50 mg/day to remain in the Treatment Period.
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 8 | 10
percentage of change from baseline score
  Visit 3 | -17.06 (9.47) | -3.50 (23.71)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | -17.93 (10.63) | -8.93 (22.95)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | -12.63 (12.24) | 1.48 (17.32)
  Visit 6: number analyzed (Participants) | 6 | 6
  Visit 6 | -5.05 (20.99) | -4.99 (19.04)

5. Secondary Outcome: Number of Headache Days
Description: Number of Headache Days reported in 30-day Baseline Period and Treatment Period Months 1-12
Time Frame: Baseline and Months 1-12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Headache days
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 10 | 10
Headache days
  Baseline | 22.95 (4.39) | 23.77 (4.64)
  Month 1: number analyzed (Participants) | 9 | 10
  Month 1 | 18.41 (5.96) | 21.67 (4.28)
  Month 2: number analyzed (Participants) | 8 | 10
  Month 2 | 16.50 (7.61) | 17.54 (6.81)
  Month 3: number analyzed (Participants) | 8 | 10
  Month 3 | 16.83 (7.12) | 18.37 (7.76)
  Month 4: number analyzed (Participants) | 8 | 9
  Month 4 | 15.74 (8.09) | 14.39 (10.05)
  Month 5: number analyzed (Participants) | 6 | 9
  Month 5 | 11.34 (7.17) | 13.47 (8.95)
  Month 6: number analyzed (Participants) | 6 | 9
  Month 6 | 15.18 (6.07) | 16.58 (7.68)
  Month 7: number analyzed (Participants) | 6 | 8
  Month 7 | 12.64 (6.39) | 12.54 (9.23)
  Month 8: number analyzed (Participants) | 6 | 6
  Month 8 | 12.36 (5.16) | 11.5 (7.26)
  Month 9: number analyzed (Participants) | 6 | 6
  Month 9 | 12.02 (5.6) | 9.96 (5.71)
  Month 10: number analyzed (Participants) | 6 | 5
  Month 10 | 6.93 (4.59) | 8.02 (1.06)
  Month 11: number analyzed (Participants) | 5 | 5
  Month 11 | 8.36 (6.5) | 8.51 (6.09)
  Month 12: number analyzed (Participants) | 5 | 5
  Month 12 | 7.51 (5.04) | 8.06 (5.34)

6. Secondary Outcome: Headache Impact Test (HIT-6) Scores at Visits 2-6 to Measure Effect of Headache in Subject's Life
Description: The Headache Impact Test (HIT-6) is a tool used to measure the impact headaches have on an individual's ability to function on the job, at school, at home and in social situations. The HIT-6 score range is from 36 to 78 with higher scores indicating greater impact (worse outcome).
Time Frame: Collected on Visit 2 (Day 29), 3 (Day 113), Visit 4 (Day 197), Visit 5 (281), and Visit 6 (Day 365)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Visit 2 | 66.40 (5.19) | 66.50 (3.84)
  Visit 3: number analyzed (Participants) | 9 | 10
  Visit 3 | 61.89 (6.92) | 59.9 (7.77)
  Visit 4: number analyzed (Participants) | 6 | 10
  Visit 4 | 54.5 (5.39) | 60.44 (8.19)
  Visit 5: number analyzed (Participants) | 6 | 9
  Visit 5 | 52.83 (7.44) | 58.71 (7.85)
  Visit 6: number analyzed (Participants) | 6 | 7
  Visit 6 | 52.57 (7.20) | 54.17 (9.81)

7. Secondary Outcome: MEWT Simple Reaction Time Sub-test Score Percent Change Compared From Baseline to Visits 3-6
Description: The Mental Efficiency Workload Test (MEWT) is a cognitive functioning scale with four sub-scales (Simple Reaction Time, Running Memory Continuous Performance Task, Matching to Sample, and Mathematical Processing). Each sub-scale has a minimum and maximum values of 1 to 10, 1 indicates the poorest level and 10 indicates the best level of cognitive functioning. MEWT sub-scale score percent change from baseline will be reported. Positive change scores represent better cognitive functioning compared to baseline.
Time Frame: Baseline, Visit 3 (Day 113), Visit 4 (Day 197), Visit 5 (281), and Visit 6 (Day 365)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline score
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 8 | 10
percentage of change from baseline score
  Visit 3 | -8.90 (18.62) | 14.22 (30.32)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | -3.20 (17.15) | 4.76 (8.44)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | -3.87 (25.48) | -4.17 (10.05)
  Visit 6: number analyzed (Participants) | 6 | 6
  Visit 6 | -3.16 (24.15) | 2.31 (18.86)

8. Secondary Outcome: MEWT Running Memory Continuous Performance Task Sub-test Score Percent Change Compared From Baseline to Visits 3-6
Description: as for outcome 7
Time Frame: Baseline, Visit 3 (Day 113), Visit 4 (Day 197), Visit 5 (281), and Visit 6 (Day 365)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline score
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 8 | 10
percentage of change from baseline score
  Visit 3 | -15.66 (38.87) | 1.13 (24.70)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | -1.20 (41.31) | 4.39 (16.55)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | -3.96 (43.64) | 18.81 (28.45)
  Visit 6: number analyzed (Participants) | 6 | 6
  Visit 6 | -6.99 (43.50) | 2.2 (31.91)

9. Secondary Outcome: MEWT Matching to Sample Sub-test Score Percent Change Compared From Baseline to Visits 3-6
Description: as for outcome 7
Time Frame: Baseline, Visit 3 (Day 113), Visit 4 (Day 197), Visit 5 (281), and Visit 6 (Day 365)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline score
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 8 | 10
percentage of change from baseline score
  Visit 3 | 19.06 (44.13) | 21.74 (27.86)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | 15.04 (47.59) | 8.59 (25.34)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | 18.49 (45.11) | 12.72 (23.34)
  Visit 6: number analyzed (Participants) | 6 | 6
  Visit 6 | 40.86 (42.88) | 24.75 (49.32)

10. Secondary Outcome: MEWT Mathematical Processing Sub-test Score Percent Change Compared From Baseline to Visits 3-6
Description: as for outcome 7
Time Frame: Baseline, Visit 3 (Day 113), Visit 4 (Day 197), Visit 5 (281), and Visit 6 (Day 365)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline score
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 8 | 10
percentage of change from baseline score
  Visit 3 | -11.23 (22.61) | 17.74 (50.54)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | -22.90 (16.48) | 16.43 (35.88)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | -23.81 (16.26) | 28.61 (48.44)
  Visit 6: number analyzed (Participants) | 6 | 6
  Visit 6 | 1.52 (8.91) | 29.44 (50.47)

11. Secondary Outcome: Subject Estimation of Compliance With Daily Study Drug
Description: Subject estimation of compliance with daily study drug during the study period. Compliance ranges from 0% to 100% with higher percentages indicating greater compliance with study drug.
Time Frame: Collected on Visit 2 (Day 29), 3 (Day 113), Visit 4 (Day 197), and Visit 5 (281)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of compliance
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 9 | 10
percentage of compliance
  Visit 2 | 100 (0) | 99.73 (0.58)
  Visit 3: number analyzed (Participants) | 8 | 10
  Visit 3 | 99.84 (0.46) | 99.73 (0.56)
  Visit 4: number analyzed (Participants) | 6 | 9
  Visit 4 | 99.55 (1.10) | 97.65 (3.09)
  Visit 5: number analyzed (Participants) | 6 | 6
  Visit 5 | 98.69 (1.61) | 99.63 (2.35)

12. Secondary Outcome: Number of Non-Serious Adverse Events Between Groups
Time Frame: 13 Months (Visit 1 to Visit 6)
Population: All consenting participants.
Measure: Mean (Standard Deviation); unit: Adverse Events
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 10 | 10
Adverse Events | 8.60 (8.93) | 4.60 (3.17)

13. Secondary Outcome: Subject's Migraine Specific Quality of Life Questionnaire (MSQ) Scores at Baseline, 3, 6, 9 and 12 Months to Measure Subject's Quality of Life
Description: The Migraine-Specific Quality of Life Questionnaire (MSQ) is a scale that measures the impact of migraine across three aspects: role function-restrictive (RR), role function-preventive (RP), and emotional function (EF). Possible scores on each sub-scale range from a 0 to 100 scale such that higher scores indicate better quality of life.
Time Frame: Baseline, Months: 3, 6, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Role Function-Restrictive - Baseline | 32.14 (16.62) | 29.71 (14.77)
  Role Function-Restrictive - Month 3: number analyzed (Participants) | 9 | 10
  Role Function-Restrictive - Month 3 | 56.51 (25.18) | 56.29 (25.16)
  Role Function-Restrictive - Month 6: number analyzed (Participants) | 6 | 9
  Role Function-Restrictive - Month 6 | 77.14 (10.22) | 59.37 (21.94)
  Role Function-Restrictive - Month 9: number analyzed (Participants) | 6 | 7
  Role Function-Restrictive - Month 9 | 79.52 (13.21) | 60.41 (25.52)
  Role Function-Restrictive - Month 12: number analyzed (Participants) | 6 | 6
  Role Function-Restrictive - Month 12 | 81.90 (12.21) | 72.38 (24.36)
  Role Function-Preventive - Baseline | 56.50 (22.61) | 46.50 (24.39)
  Role Function-Preventive - Month 3: number analyzed (Participants) | 9 | 10
  Role Function-Preventive - Month 3 | 72.78 (26.82) | 65.00 (28.28)
  Role Function-Preventive - Month 6: number analyzed (Participants) | 6 | 9
  Role Function-Preventive - Month 6 | 90.00 (8.37) | 72.22 (26.94)
  Role Function-Preventive - Month 9: number analyzed (Participants) | 6 | 7
  Role Function-Preventive - Month 9 | 88.33 (8.16) | 72.86 (26.28)
  Role Function-Preventive - Month 12: number analyzed (Participants) | 6 | 6
  Role Function-Preventive - Month 12 | 96.67 (2.58) | 80.83 (24.98)
  Emotional Function - Baseline | 39.33 (30.70) | 22.67 (22.04)
  Emotional Function - Month 3: number analyzed (Participants) | 9 | 10
  Emotional Function - Month 3 | 57.78 (36.67) | 56.67 (33.15)
  Emotional Function - Month 6: number analyzed (Participants) | 6 | 9
  Emotional Function - Month 6 | 88.89 (6.89) | 56.30 (32.51)
  Emotional Function - Month 9: number analyzed (Participants) | 6 | 7
  Emotional Function - Month 9 | 92.22 (16.01) | 70.48 (29.02)
  Emotional Function - Month 12: number analyzed (Participants) | 6 | 6
  Emotional Function - Month 12 | 95.56 (8.07) | 78.89 (28.10)

ADVERSE EVENTS:
Arm/Group | OnabotulinumtoxinA + Topiramate | OnabotulinumtoxinA + Placebo
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OnabotulinumtoxinA + Topiramate (N=10) | OnabotulinumtoxinA + Placebo (N=10)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rectal Proplapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OnabotulinumtoxinA + Topiramate (N=10) | OnabotulinumtoxinA + Placebo (N=10)
Decreased Cognition (Nervous system disorders) | 5 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Vertigo (General disorders) | 2 (3) | 4 (5)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No